CLINICAL TRIAL: NCT02152696
Title: Optimal Treatment for Women With a Persisting Pregnancy of Unknown Location - a Randomized Clinical Trial of Women at Risk for an Ectopic Pregnancy: Active Treatment Versus No Treatment
Brief Title: Optimal Treatment for Women With a Persisting Pregnancy of Unknown Location
Acronym: ACTorNOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Augusta University (Other); Penn State University (Other); University of California, San Francisco (Other); University of North Carolina (Other); University of Oklahoma (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000023590; 2U10HD055925-06 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-06-02 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-11

CONDITIONS: Persistent Pregnancy of Unknown Location; Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Expectant Management (Active Comparator): Subjects will have their PPUL expectantly managed using serum hCG monitoring.
  Interventions: Other: Expectant Management
- Uterine evacuation with MTX for some (Active Comparator): Subjects will undergo a uterine evacuation. If hCG levels do not sufficiently decrease after the uterine evacuation, the subject will be treated with methotrexate. If hCG levels do sufficiently decrease after the uterine evacuation, no further treatment is required.
  Interventions: Drug: Methotrexate; Procedure: Uterine Evacuation
- Empiric treatment with MTX for all (Active Comparator): Subjects will be treated with methotrexate, receiving one dose on day 0 and a subsequent dose on day 4. Additional doses will be administered as needed based on hCG levels.
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — Two Dose Protocol: The patient will receive the first dose of MTX 50mg/m2 on treatment day 0. She will receive a second dose of MTX 50mg/m2 on treatment day 4 and a serum hCG level will be drawn. Subsequent doses of MTX will be administered based on hCG levels.
  Arms: Empiric treatment with MTX for all; Uterine evacuation with MTX for some
Procedure: Uterine Evacuation — Uterine evacuation or dilation and curettage. At the clinician's discretion, this can be performed using local anesthesia, sedation or general anesthesia and can use a manual or electrical evacuation.
  Arms: Uterine evacuation with MTX for some
Other: Expectant Management — Pregnancy will be expectantly managed using serum hcg monitoring
  Arms: Expectant Management

SUMMARY:
This is a randomized controlled trial to compare three currently available management strategies for women with a persisting pregnancy of unknown location (PPUL), which makes them at-risk for ectopic pregnancy. We will recruit hemodynamically stable women with a confirmed PPUL to be randomized to one of three strategies: 1) Uterine evacuation followed by methotrexate (MTX) for some (those that have evidence of a non visualized ectopic pregnancy) 2) Empiric treatment with MTX for all 3) Expectant management. Randomization will be 1:1:1 into these three arms. After randomization, they will be followed and treated clinically as is indicated by the progression of their condition. Primary outcome measures: uneventful decline of hCG to 5 IU/mL.

ELIGIBILITY:
Inclusion Criteria:

* Female with a persisting pregnancy of unknown location:
* A pregnancy of unknown location is defined as a pregnancy in a woman with a positive pregnancy test but no definitive signs of pregnancy in the uterus or adnexa on ultrasound imaging. A definitive sign of gestation includes ultrasound visualization of a gestational sac with a yolk sac (with or without an embryo) in the uterus or in the adnexa. Ultrasound must be performed within 7 days prior to randomization.
* Persistence of hCG is defined as at least 2 serial hCG values (over 2-14 days), showing < 15% rise per day, or < 50% fall between the first and last value.
* Patient is hemodynamically stable, hemoglobin >10 mg/dL
* Greater than or 18 years of age

Exclusion Criteria:

* Hemodynamically unstable in need of acute treatment
* Most recent hCG > 5000 mIU/mL
* Patient obtaining care in relation to a recently completed pregnancy (delivery, spontaneous or elective abortion)
* Diagnosis of gestational trophoblastic disease
* Subject unwilling or unable to comply with study procedures
* Known hypersensitivity to MTX
* Presence of clinical contraindications for treatment with MTX
* Prior medical or surgical management of this gestation
* Subject unwilling to accept a blood transfusion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2014-07-25 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esther Eisenberg, MD MPH, Study Director — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD); Nanette Santoro, MD, Study Chair — University of Colorado, Denver; Kurt Barnhart, MD MSCE, Principal Investigator — University of Pennsylvania; Michael Diamond, MD, Study Director — Augusta University; Richard Legro, MD, Study Director — Penn State University; Marcelle Cedars, MD, Study Director — University of California, San Francisco; Anne Steiner, MD MPH, Study Director — University of North Carolina; Karl Hansen, MD PhD, Study Director — University of Oklahoma; Christos Coutifaris, MD PhD, Study Director — University of Pennsylvania; Heping Zhang, PhD, Study Director — Yale University
Locations (17):
- United States (17):
  - University of California San Francisco, San Francisco, California
  - Denver Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of South Florida, Tampa, Florida
  - Augusta University, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - University Of Illinois at Chicago, Chicago, Illinois
  - Wayne State University, Southfield, Michigan
  - Washington University, St Louis, Missouri
  - University of Rochester, Rochester, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Carolinas Medical Center - Women's Institute, Charlotte, North Carolina
  - Duke University, Durham, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville, South Carolina
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other researchers through the NICHD DASH system. It will be available 6 months after publication of the primary results.

REFERENCES:
- [Derived] Barnhart KT, Hansen KR, Stephenson MD, Usadi R, Steiner AZ, Cedars MI, Jungheim ES, Hoeger KM, Krawetz SA, Mills B, Alston M, Coutifaris C, Senapati S, Sonalkar S, Diamond MP, Wild RA, Rosen M, Sammel MD, Santoro N, Eisenberg E, Huang H, Zhang H; Reproductive Medicine Network. Effect of an Active vs Expectant Management Strategy on Successful Resolution of Pregnancy Among Patients With a Persisting Pregnancy of Unknown Location: The ACT or NOT Randomized Clinical Trial. JAMA. 2021 Aug 3;326(5):390-400. doi: 10.1001/jama.2021.10767. PMID 34342619

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Expectant Management | Uterine Evacuation With MTX for Some | Empiric Treatment With MTX for All
Started | 86 | 87 | 82
Completed | 86 | 86 | 81
Not Completed | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Expectant Management | Uterine Evacuation With MTX for Some | Empiric Treatment With MTX for All | Total
Number analyzed (Participants) | 86 | 87 | 82 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.1 (5.6) | 31.2 (5.9) | 31.5 (5.7) | 31.6 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86 | 87 | 82 | 255
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 6 | 17
  Not Hispanic or Latino | 80 | 75 | 74 | 229
  Unknown or Not Reported | 3 | 4 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 10 | 4 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 37 | 33 | 32 | 102
  White | 41 | 40 | 39 | 120
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 7 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 87 | 82 | 255
Estimated gestational age - week [Mean (Standard Deviation); unit: weeks] — Population: Data were missing for 1 patient in the Expectant management group, 4 in the Uterine evacuation with MTX for some group and 2 in the Empiric treatment with MTX for all.
  weeks
    number analyzed (Participants) | 85 | 83 | 80 | 248
    (all) | 6.4 (1.8) | 6.9 (1.9) | 6.7 (2.0) | 6.7 (1.9)
First hCG value at screening (mIU/ml) [Mean (Standard Deviation); unit: mIU/ml] | 661.2 (688.6) | 561.9 (702.5) | 633.3 (695.8) | 618.3 (694.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Uneventful Clinical Resolution of a Pregnancy of Unknown Location Without Change From the Initial Management Strategy
Description: The primary outcome measure in each of each 3 treatment arm is the uneventful clinical resolution of a PPUL without change in treatment from the initial management strategy.
Time Frame: 6 weeks from randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Expectant Management | Uterine Evacuation With MTX for Some | Empiric Treatment With MTX for All
Number analyzed (Participants) | 86 | 87 | 82
Participants | 31 | 42 | 45

ADVERSE EVENTS:
Time Frame: The period of time over which the adverse events were collected is: from the initiation of the study procedures to the end of the study treatment follow-up, which is about an average of 42 days following the last administration of study treatment.
Arm/Group | Expectant Management | Uterine Evacuation With MTX for Some | Empiric Treatment With MTX for All
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/87 | 0/82
Serious Adverse Events (participants affected / at risk) | 2/86 | 2/87 | 0/82
Other Adverse Events (participants affected / at risk) | 44/86 | 53/87 | 46/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Management (N=86) | Uterine Evacuation With MTX for Some (N=87) | Empiric Treatment With MTX for All (N=82)
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) — Hospitalization.ED visit pelvic ultrasound revealed right adnexal mass concerning for tubal pregnancy.
Salpingectomy (Pregnancy, puerperium and perinatal conditions) | 2 | 0 (0) | 0 (0)
Right ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Expectant Management (N=86) | Uterine Evacuation With MTX for Some (N=87) | Empiric Treatment With MTX for All (N=82)
One or more adverse event (General disorders) | 44 (44) | 53 (53) | 46 (46)
Nausea (Gastrointestinal disorders) | 22 (22) | 32 (32) | 31 (31)
Vomiting (Gastrointestinal disorders) | 2 (2) | 11 (11) | 10 (10)
Pelvic Pain (Reproductive system and breast disorders) | 37 (37) | 42 (42) | 38 (38)
Loss of Appetite (Gastrointestinal disorders) | 25 (25) | 28 (28) | 23 (23)
Mouth Sores (Gastrointestinal disorders) | 5 (5) | 6 (6) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 9 (9) | 21 (21) | 13 (13)
Heart Burn/Indigestion (General disorders) | 7 (7) | 12 (12) | 5 (5)
Hair Loss (General disorders) | 4 (4) | 9 (9) | 6 (6)
Headaches (Nervous system disorders) | 31 (31) | 25 (25) | 27 (27)
Fatigue (General disorders) | 38 (38) | 38 (38) | 36 (36)
Vaginal bleeding (Surgical and medical procedures) | 38 (38) | 46 (46) | 39 (39)
Dizziness or weakness (General disorders) | 18 (18) | 27 (27) | 17 (17)
Shoulder or back pain (General disorders) | 14 (14) | 18 (18) | 12 (12)
Persistent dry cough (General disorders) | 3 (3) | 5 (5) | 5 (5)
Any Other Side Effects (General disorders) | 6 (6) | 4 (4) | 3 (3) — Including sore throats, cough, constipation, depression, lower back pain, pain in breasts/shoulder, and other unspecified events. These events were recorded in free text, not separated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT02152696/Prot_SAP_000.pdf